CLINICAL TRIAL: NCT04086498
Title: Effects of Ketonemia and Glycemia Variations During Ketogenic and Mediterranean Weight Loss Diets on Appetite Levels, Executive Functions and Mood
Brief Title: Effects of a Ketogenic Diet on Psychological Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Antonio Paoli, Professor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: KDPSY2
Record Dates: First submitted 2019-08-29; First posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Overweight; Mood; Appetitive Behavior
Keywords: ketogenic diet; Mediterranean diet; ketones; glycaemia; executive functions
MeSH Terms: conditions — Overweight; Appetitive Behavior; Ketosis | interventions — Diet, Mediterranean

STUDY DESIGN:
Intervention Model Description: It is single blind, parallel arms study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Raw data are encoded with 3 letters assigned to each treatment (A, B and C). Investigators and outcomes assessor do not have access to the waiting (letter-treatment)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ketogenic-mediterranean diet with phytoextracts (Experimental): The KEMEPHY diet (Paoli et al., 2011) is a mediterranean calorie-controlled ketogenic protocol (about 900 Kcal/day) with the use of some phytoextracts. During this protocol subjects are allowed to eat with no limits green leafy vegetables, cruciferous, zucchini, cucumbers and eggplants. The quantity of meat, eggs and fish was limited to once a day (120g of meat or 200g of fish or 1 egg). Moreover, subjects daily consumed four food supplements and liquid herbal extracts. Food supplements are high proteins (19g/portion) and very low carbohydrate (3.5g/portion) formulas simulating the aspect and taste of common carbohydrate rich foods added with dry phytoextracts (Lodi et al., 2016).
  Interventions: Other: KEMEPHY
- Ketogenic Diet (Active Comparator): The KD is a protocol in which all foods containing carbohydrate are excluded, whereas meat, eggs, fish, ham, green leafy vegetables, cruciferous, zucchini, cucumbers and eggplants can be eat without any limit. This protocol allows the use of oil, lemon juice (2 tbs/day), spices and aromatic herbs with a limitation of the use of saturated fats like butter, margarine and lard. Coffee, tea and herbal tea could be sweetened with sweeteners
  Interventions: Other: KD
- Mediterranean Diet (Active Comparator): The MD is a balanced calorie-controlled diet. The calorie intake was 1200 Kcal/day of which 15% were proteins, 60% carbohydrates and 25% fat. In this protocol was highlighted the use of the typical ingredients of the mediterranean tradition, such as extravirgin olive oil, vegetables, fruits, fish, lean meat and whole grain cereals.
  Interventions: Other: Mediterranean diet

INTERVENTIONS:
Other: Mediterranean diet — The group received a plan for a isocaloric Mediterranean Diet
  Arms: Mediterranean Diet
Other: KEMEPHY — The group received a plan for a ketogenic mediterranean with herbal extracts diet
  Arms: ketogenic-mediterranean diet with phytoextracts
Other: KD — The group received a plan for a low carbohydrate ketogenic diet
  Arms: Ketogenic Diet

SUMMARY:
The aim of the study is to investigate how glycemia and ketonemia variations during three different diet protocols: a ketogenic diet without any restriction on calories intake (KD), a calorie-restricted ketogenic-mediterranean diet (KEMEPHY) and a calorie-restricted mediterranean diet (MD) affect appetite, executive functions and mood in overweight young women.

DETAILED DESCRIPTION:
Fifty overweight young women with a body mass index (BMI) greater than 25 will be randomly assigned to a ten days of ketogenic diet (KD), calorie-restricted ketogenic-mediterranean diet (KEMEPHY) or Mediterranean diet (MD). All subjects will begin the prescribed diet at the beginning of their follicular phase. Body composition, fasting blood glucose and β-hydroxybutyrate (BHB), visual analogue scale (VAS) to test appetite as well as psychological tests (one mood test and two cognitive tasks) will be obtained 5 days before the beginning and on the last day of the diet-period.

ELIGIBILITY:
Inclusion Criteria:

* female sex age between 20 and 35 years,
* 25<BMI>39.9 kg/m2

Exclusion Criteria:

* smokers,
* subjects under diet-treatment,
* subjects treated for diseases such as diabetes,
* cardiovascular diseases,
* depression,
* subjects doing sport more than 2 hours per week.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2016-06-15 (Actual)

PRIMARY OUTCOMES:
Motivation to eat and appetite | after 8 weeks
  Motivation to eat and appetite were investigated by Visual Analog Scale (Hill & Blundell, 1982) , a test formed by 6 scales. Each scale was 10 cm long and was labelled with vertical lines and numbers (from 0 to10) every cm. Participants had to choose which part of the scale better described how they felt. The scale investigated appetite, fullness, desire to eat, how much would participant eat, urgency of eating and worries about food through 6 questions. Moreover, also the unfullness index (10 - fullness) was taken into account (R. J. Stubbs et al., 2000).
cognitive task1 | after 8 weeks
  The working memory test was an adapted version of the visuo-spatial N-back (Cui, Bray, Bryant, Glover, & Reiss, 2011; Haberecht et al., 2001). It consisted in remembering the position of the letter "o" that, in each trial, could appear in different positions, since a 9-part grid divides the screen. Number of correct or incorrect answers will be counted
Cognitive task2 | after 8 weeks
  The executive function test was an adapted version of the inhibitory control task (Amodio et al., 2010; Cona, Arcara, Amodio, Schiff, & Bisiacchi, 2013) . The stimulus were letters that appear in the centre of the screen. The task was formed by two main parts. In the first one the participant had to respond when the letter x or y appeared on the screen; in the second part the participant had to answer only when x preceded y and then vice versa. Number of correct or incorrect answers will be counted

SECONDARY OUTCOMES:
body water content | after 8 weeks
  Body composition will be assessed by body electrical impedance analysis (BIA) that measures Total body water and intra and extracellular water in liters
lean body mass | after 8 weeks
  Body composition will be assessed by body electrical impedance analysis (BIA) that measures lean body mass in kg
fat body mass | after 8 weeks
  Body composition will be assessed by body electrical impedance analysis (BIA) that measures fat body mass in kg
Mood | after 8 weeks
  The mood test was the Italian Version of the Depression Anxiety Stress Scales-21. It was a self report measure formed by 21 items that reliably measure depression (lack of incentive, dysphoria and low self-esteem) as well as anxiety (somatic and subjective symptoms), stress (irritability, impatience, tension and arousal) and general distress (related to anxiety and depression) (Bottesi et al., 2015). The responses are given on a 4-point Likert scale, ranging from zero if "I strongly disagree" to 3 if "I totally agree".
blood glucose | after 8 weeks
  to assess diets' effects on glycaemia, capillary blood will be analyzed. We measure glucose in mg/100ml
blood ketones | after 8 weeks
  to assess diets' effects on ketonemia, capillary blood will be analyzed. We measure ketone in mol/L

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Paoli, MD, Principal Investigator — University of Padova
Locations (1):
- Nutrition and Exercise Lab, DSB, University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Raw data of measured variables

REFERENCES:
- [Background] Lodi A, Karsten B, Bosco G, Gomez-Lopez M, Brandao PP, Bianco A, Paoli A. The Effects of Different High-Protein Low-Carbohydrates Proprietary Foods on Blood Sugar in Healthy Subjects. J Med Food. 2016 Nov;19(11):1085-1095. doi: 10.1089/jmf.2016.0072. Epub 2016 Oct 18. PMID 27754766
- [Background] Paoli A, Bosco G, Camporesi EM, Mangar D. Ketosis, ketogenic diet and food intake control: a complex relationship. Front Psychol. 2015 Feb 2;6:27. doi: 10.3389/fpsyg.2015.00027. eCollection 2015. PMID 25698989
- [Background] Paoli A. Ketogenic diet for obesity: friend or foe? Int J Environ Res Public Health. 2014 Feb 19;11(2):2092-107. doi: 10.3390/ijerph110202092. PMID 24557522
- [Background] Paoli A, Bianco A, Grimaldi KA, Lodi A, Bosco G. Long term successful weight loss with a combination biphasic ketogenic Mediterranean diet and Mediterranean diet maintenance protocol. Nutrients. 2013 Dec 18;5(12):5205-17. doi: 10.3390/nu5125205. PMID 24352095
- [Background] Paoli A. Booster Ketones: Battling Hunger. Obesity (Silver Spring). 2018 Feb;26(2):252-253. doi: 10.1002/oby.22099. Epub 2018 Jan 10. No abstract available. PMID 29318785
- [Background] Stubbs BJ, Cox PJ, Evans RD, Cyranka M, Clarke K, de Wet H. A Ketone Ester Drink Lowers Human Ghrelin and Appetite. Obesity (Silver Spring). 2018 Feb;26(2):269-273. doi: 10.1002/oby.22051. Epub 2017 Nov 6. PMID 29105987